CLINICAL TRIAL: NCT07237685
Title: Evaluating Atherosclerotic Disease Progression in High-Risk Patients With Diabetes Mellitus
Brief Title: Evaluating Atherosclerotic Disease Progression in Patients With Diabetes Mellitus
Acronym: EVOLVE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Horizon Innovative Health Initiative (Unknown); Novo Nordisk A/S (Industry); INSTITUTO DE INVESTIGACION BIOMEDICA DE SALAMANCA (IBSAL) (Unknown); Cardiology Centers of the Netherlands (Unknown)
Responsible Party: Principal Investigator, M.M. Winter, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: NL86138.018.24
Record Dates: First submitted 2025-09-24; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease (CAD); Atherosclerosis Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
People with type 2 diabetes have a much higher risk of heart disease. One common problem is when the blood vessels that supply the heart become narrowed or blocked by fatty deposits, called plaque. This makes it harder for blood to reach the heart and can lead to serious problems such as chest pain, heart attacks, or even death.

This study will follow people with type 2 diabetes who have already had a special heart scan called a coronary CT angiography. This scan takes detailed pictures of the heart's blood vessels.

The goal is to understand how heart disease changes over time in people with type 2 diabetes, by looking at repeat scans and other health information. By learning more about how plaque builds up or gets worse, researchers hope to find better ways to identify which patients are most at risk for future heart problems.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Previous completion of CCTA scan for CAD assessment
* Diagnosed with Type 2 Diabetes and currently receiving glucose lowering treatment
* Sufficient image quality of the CCTA scan (at least 2/3 vessels of sufficient quality for assessment).

Exclusion Criteria:

* Inability to provide written informed consent
* Presence of an unstable condition
* Ingeligibility for CCTA acquisition due to severe renal dysfunction (eGFR ≤ 30 mL/min/1.73m²) or known hypersensitivity or contraindication to CT contrast agents
* Any other treatment or clinically relevant condition that could interfere with the conduct or interpretation of the study in the opinion of the investigator
* inability or unwillingness to comply with the protocol requirements, or deemed by investigator to be unfit for the study
* Baseline (routine care) CCTA performed < 2 years or > 5 years before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, patients with T2D who previously undergone CCTA for CAD assessment will be recruited. Patients will be included at three clinical sites: Amsterdam UMC, Cardiology centre Netherlands (CCN), University hospital of Salamanca - Fundacion Instituto de Estudios de ciencias de la salud de castilla y leon (IBSAL).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2036-10-01 (Estimated)

PRIMARY OUTCOMES:
progression of total coronary plaque volume (mm3) | Between baseline (retrospective) and follow up CCTA (interval 2-5 years).
  The primary study parameter will be the progression of total coronary plaque volume (mm3). This will be calculated by subtracting the coronary plaque volume measured in the first CCTA from the total plaque volume measured in the follow-up CCTA. The plaque volume will be determined by dividing the total plaque volume by the total vesssel volume

SECONDARY OUTCOMES:
Changes in Coronary Artery Disease Reporting and Data Scale(CAD-RADS) scores | Between baseline (retrospective) and follow up CCTA (interval 2-5 years)
  Change in the percentage of luminal narrowing per lesion as defined by the Coronary Artery Disease Reporting and Data Scale(CAD-RADS) score (minimum 0, maximum 5).
Progression of calcified plaque volume (mm3) | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  The progression of total calcified plaque volume
Progression of non-calcified plaque volume (mm3) | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  The progression of total non-calcified plaque volume
Progression of low attenuation plaque volume (mm3) | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  The progresison of total low attenuation plaque volume
Changes in coronary artery calcium score | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  Change in the coronary artery calcium score
Changes in the number of high-risk plaque characteristics | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  * Spotty calcium defined as punctate calcium within a plaque
  * Napkin ring sign defined in a non-calcified plaque cross sectional image by the presence of two or more features: a central area of low attenuation plaque that is apparently in contact with the lumen; and a ring like peripheral rim of higher CT attenuation surrounding his central area.
  * Positive remodeling, defined as the ratio of outer vessel diameter at the site of plaque divided by the average outer diameter of the proximal and distal vessel greater than 1.1.
  * Low attenuation plaque, defined as non-calcified plaque with internal attenuation less than 30 Hounsfield units (HU).
Changes in peri coronary fat attenuation index | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  Change in the peri coronary fat attenuation index
The number of cardiovascular events | Baseline (retrospective) and follow up CCTA (interval 2-5 years)
  The number of cardiovascular events consisting of:
  * Myocardial infarction (defined as the universal definition as established by the European Society of Cardiology (ESC), American College of Cardiology (ACC), American Heart Association (AHA) and the World health federation)
  * Cerebrovascular accidents (neurologic deficit lasting more than 24 hours or lasting less than 24 hours with a brain imaging study showing infarction)
  * Target vessel revascularization
  * CAD related hospitalization
The number of cardiovascular events | Baseline CCTA untill 10 years follow up after inclusion
  Myocardial infarction (defined as the universal definition as established by the European Society of Cardiology (ESC), American College of Cardiology (ACC), American Heart Association (AHA) and the World health federation)
  * Cerebrovascular accidents (neurologic deficit lasting more than 24 hours or lasting less than 24 hours with a brain imaging study showing infarction)
  * Target vessel revascularization
  * CAD related hospitalization

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam University Medical Centers, Amsterdam
  - Cardiology Centers of the Netherlands, Amsterdam